CLINICAL TRIAL: NCT06870461
Title: Hepatic Excision and Ablation Log
Acronym: HEAL
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Other Study IDs: 003810
Record Dates: First submitted 2024-12-18; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-03

CONDITIONS: Malignant Liver Tumor; Benign Liver Tumor
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Liver surgery / ablation — Any type of liversurgery or CT-guidede liver ablation

SUMMARY:
This study aims to establish a registry for liver surgery and ablation procedures to improve patient care, advance research, and enhance surgical quality. The registry will collect pseudonymized data on patient demographics, disease characteristics, procedural details, and outcomes.

DETAILED DESCRIPTION:
The purpose of this registry is to create a comprehensive list of individuals who have undergone liver surgery or liver ablation, allowing researchers and clinicians to assess their data in future studies if they meet the eligibility criteria. All patients who have received liver surgery or liver ablation procedures at our institution will be included in this registry.

Information collected as part of the registry will be used solely to assess potential participants' eligibility for research studies, allowing for the evaluation of long-term outcomes, identification of risk factors, and investigation of therapeutic interventions. This data will help to enhance the understanding of the patient population undergoing liver surgery and improve clinical practices.

A patient registry is an organized system that uses observational study methods to collect standardized clinical data and other relevant information. It aims to evaluate specific outcomes for individuals who have undergone liver surgery or ablation, serving scientific, clinical, and policy-related purposes. The registry will support the development of targeted research studies and provide valuable insights into the treatment and management of liver diseases.

ELIGIBILITY:
Inclusion Criteria:

* Both benign and malignant liver lesions are included

Exclusion Criteria:

- Intervention performed solely for liver biopsy, without any subsequent surgical resection or ablation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who will undergo liver surgery or ablation.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2035-01 (Estimated); Study Completion 2040-01 (Estimated)

PRIMARY OUTCOMES:
Establishment of a Liver Surgery and Ablation Registry | 10 years
  The primary objective of this study is to create a comprehensive registry of patients who have undergone liver surgery or liver ablation. This registry will serve as a foundation for future epidemiological studies, enabling the assessment of long-term outcomes, the identification of risk factors, and the evaluation of potential therapeutic interventions. Data collected will include demographic information, medical history, surgical details, postoperative outcomes, and survival rates. By compiling this data, we aim to better understand the patient population and improve care for individuals undergoing liver surgery or ablation.

CONTACTS AND LOCATIONS:
Overall Officials: Thiery Chapelle, Principal Investigator — University Hospital, Antwerp

IPD SHARING:
Plan to Share IPD: No